CLINICAL TRIAL: NCT01074762
Title: The Diabetes Care in General Practice Study: Randomised Controlled Trial of Structured Personal Care of Type 2 Diabetes Mellitus
Brief Title: Randomised Controlled Trial of Structured Personal Care of Type 2 Diabetes Mellitus
Acronym: DCGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Responsible Party: Niels de Fine Olivarius, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DCGP1989
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2003-07

CONDITIONS: Diabetes Mellitus; Quality of Health Care; Health Services Research
Keywords: Diabetes mellitus; Quality of health care; Health services research
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Routine general practice care (No Intervention): In the comparison group, doctors were free to choose any treatment and change it over time. The study coordinating centre did not contact comparison practices after the end of recruitment (late 1991) until 1995.
  Interventions: Behavioral: Structured personal care

INTERVENTIONS:
Behavioral: Structured personal care — General practitioners (GPs) were recommended to perform regular follow up every three months and an annual screening for diabetic complications. The GP was requested to define, together with the patient, the best possible goals for blood glucose concentration, glycated haemoglobin (HbA1c), diastolic blood pressure, and lipids within three predefined categories. At each quarterly consultation, the GP was asked to compare the achievements with the goal and consider changing either goal or treatment accordingly. The doctors received annual descriptive feedback reports on individual patients. The GPs were introduced to possible solutions to therapeutic problems through clinical guidelines supported by an annual half day seminar. Patient leaflets were produced for the doctor to hand out.

SUMMARY:
The aims of a concluding 14-year follow-up study are:

* To investigate what long-term effect the project model for structured, personalized diabetes care has on 1) the patients' mortality and development of diabetic complications, 2) the patients' use of services from the primary and secondary sector, 3) the patients' self-rated health and motivation, and 4) the doctor-patient relationship.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is an increasingly common illness that is linked to considerable excessive mortality. There are many indications that treatment of raised blood pressure and blood glucose as well as dyslipidaemia can postpone the development of diabetic complications. Treatment of T2DM is primarily done in general practice, where the results are not satisfactory. The purpose of the project is to create a basis so the existing research-based knowledge can be used to improve the quality of diabetes care in general practice.

The answer will be based on the information from 1,428 newly diagnosed diabetic patients aged 40 or over who were followed since 1989 in a randomised trial among more than 600 general practitioners. The intervention, which ended at the beginning of 1996, provided optimum conditions for follow-up, doctor-patient communication and treatment, among other ways by training the doctors, producing clinical guidelines and setting individual treatment goals. In the project, the general practitioner is seen as the coordinator of the whole health system's prophylactic efforts in relation to the individual diabetic patient.

The aims of a concluding 14-year follow-up are:

* To investigate what long-term effect the project model for structured, personalized diabetes care has on 1) the patients' mortality and development of diabetic complications, 2) the patients' use of services from the primary and secondary sector, 3) the patients' self-rated health and motivation, and 4) the doctor-patient relationship.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged 40 or older with newly diagnosed diabetes between 1 March 1989 and 28 February 1991 based on hyperglycaemic symptoms or raised blood glucose values measured in general practice

Exclusion Criteria:

* threatening somatic disease, severe mental illness, or unwillingness to participate. For our analysis, we also excluded non-white patients and patients whose diagnosis was not established by a blood glucose measurement at a major laboratory within 500 days after diagnosis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1470 (Actual)
Dates: Start 1989-03; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

PRIMARY OUTCOMES:
Mortality | From diabetes diagnosis until median14 year after study start
  The vital status of all patients was certified on the 31 January, 2006 through The Danish Civil Registration System (www.cpr.dk) which includes complete and continuously updated information on all Danish residents on vital status.
Diabetic retinopathy | at 6 year and 14 year after study start
  Incidence of diabetic retinopathy
Urinary albumin concentration | at 6 year and 14 year after study start
  Incidence of urinary albumin concentration > 15 mg/l
Myocardial infarction | From diabetes diagnosis until median14 year after study start
  Incidence of myocardial infarction. The national hospital discharge registry provided information on hospital admissions for myocardial infarction, stroke, and amputation from diagnosis until December 31, 2005.
Stroke | From diabetes diagnosis until median14 year after study start
  Incidence of stroke. The national hospital discharge registry provided information on hospital admissions for myocardial infarction, stroke, and amputation from diagnosis until December 31, 2005.

SECONDARY OUTCOMES:
New peripheral neuropathy | at 6 year and 14 year after study start
New angina pectoris | at 6 year and 14 year after study start
New intermittent claudication | at 6 year and 14 year after study start
Amputation | From diabetes diagnosis until median14 year after study start
  Incidence of amputation. The national hospital discharge registry provided information on hospital admissions for myocardial infarction, stroke, and amputation from diagnosis until December 31, 2005.

CONTACTS AND LOCATIONS:
Locations (1):
- The Research Unit for General Practice in Copenhagen, Centre for Health and Community, Øster Farimagsgade 5, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Arreskov AB, Olsen MA, Pouplier SS, Siersma V, Andersen CL, Friis S, de Fine Olivarius N. The impact of cancer on diabetes outcomes. BMC Endocr Disord. 2019 Jun 11;19(1):60. doi: 10.1186/s12902-019-0377-0. PMID 31185995
- [Derived] Heltberg A, Siersma V, Andersen JS, Ellervik C, Bronnum-Hansen H, Kragstrup J, de Fine Olivarius N. Socio-demographic determinants and effect of structured personal diabetes care: a 19-year follow-up of the randomized controlled study diabetes Care in General Practice (DCGP). BMC Endocr Disord. 2017 Dec 8;17(1):75. doi: 10.1186/s12902-017-0227-x. PMID 29216868
- [Derived] Krag MO, Hasselbalch L, Siersma V, Nielsen AB, Reventlow S, Malterud K, de Fine Olivarius N. The impact of gender on the long-term morbidity and mortality of patients with type 2 diabetes receiving structured personal care: a 13 year follow-up study. Diabetologia. 2016 Feb;59(2):275-85. doi: 10.1007/s00125-015-3804-4. Epub 2015 Nov 26. PMID 26607637
- [Derived] Larsen JR, Siersma VD, Davidsen AS, Waldorff FB, Reventlow S, de Fine Olivarius N. The excess mortality of patients with diabetes and concurrent psychiatric illness is markedly reduced by structured personal diabetes care: A 19-year follow up of the randomized controlled study Diabetes Care in General Practice (DCGP). Gen Hosp Psychiatry. 2016 Jan-Feb;38:42-52. doi: 10.1016/j.genhosppsych.2015.10.001. Epub 2015 Oct 19. PMID 26602087
- [Derived] Lundstrom H, Siersma V, Nielsen AB, Brodersen J, Reventlow S, Andersen PK, de Fine Olivarius N. The effectiveness of structured personal care of type 2 diabetes on recurrent outcomes: a 19 year follow-up of the study Diabetes Care in General Practice (DCGP). Diabetologia. 2014 Jun;57(6):1119-23. doi: 10.1007/s00125-014-3204-1. Epub 2014 Mar 6. PMID 24599111
- [Derived] Hansen LJ, Siersma V, Beck-Nielsen H, de Fine Olivarius N. Structured personal care of type 2 diabetes: a 19 year follow-up of the study Diabetes Care in General Practice (DCGP). Diabetologia. 2013 Jun;56(6):1243-53. doi: 10.1007/s00125-013-2893-1. Epub 2013 Apr 3. PMID 23549519